CLINICAL TRIAL: NCT06311357
Title: Effects of Body Weight Change in the Medical Supplement Group in Patients with Early Breast Cancer During Chemotherapy: a Randomized, Controlled Trial
Brief Title: Percent Weight Change in the Medical Supplement Group of Early Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 100/2566
Record Dates: First submitted 2023-12-12; First posted 2024-03-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-03

CONDITIONS: Early Stage Breast Cancer
Keywords: Medical supplement; Weight change in early breast cancer treatment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Nutritional advise
- Intervention (Experimental): Medical supplement and nutritional advise
  Interventions: Dietary Supplement: Ensure

INTERVENTIONS:
Dietary Supplement: Ensure — Ensure 6 scoops dietary supplement powder in 250 ml of water, 2 drinks per days for 12 weeks.
  Arms: Intervention

SUMMARY:
The goal of this RCT is to compare percent weight change in early breast cancer who takes medical supplement or not, during treatment with chemotherapy (standard AC regimen).

The main question is

• the change of weight (%) before and after complete treatment of breast cancer therapy.

Participants will be randomized into 2 group

* intervention group - receive medical supplement daily during chemotherapy treatment.
* control group - Nutritional advise during chemotherapy treatment.

DETAILED DESCRIPTION:
1. The rational is to prove the hypothesis is that, the effect of medical supplement with nutritional advise can prevent the reduction of body weight, malnutrition and treatment complication, which eventually to improve of the quality of life.
2. Primary endpoint of the study is to compare the effect of medical supplement on percent weight change in early breast cancer who received chemotherapy in Rajavithi hospital. Secondary endpoints are nutritional status (PG-SGA), quality of life.
3. Sample size formula based on Bernard R. Fundamentals of biostatistics. 5th ed. Duxbery: Thomson learning; 2000. Enrollment of 40 patients.
4. Randomization into 2 groups. Intervention arm : receive medical supplement daily (1 drink = 6 scoops in 250 ml water, 2 drinks/day) with nutritional advise. Control arm : nutritional advise only. Duration of treatment is 12 weeks
5. Enrollment and data monitoring is assessed by the staffs of oncology department in Rajavithi hospital and the data will be recorded in computer based information system.
6. Data assessment on week 0,6,12 during chemotherapy treatment.
7. Data analyzed by descriptive statistics to characterize patients at entry. We did the efficacy analyses with intention to treat population
8. We did analyses with R version 3.3.0.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological confirmed diagnosis of breast cancer
* Breast cancer stage I-III
* Recieve adjuvant or neoadjuvant doxorubicin and cyclophosphamide at Rajavithi hospital
* LVEF >= 60% - ECOG score 0-1

Exclusion Criteria:

* No indication for chemotherapy
* Contraindication for chemotherapy
* Breast cancer stage IV
* Diabetic mellitus who requires insulin injection
* BMI >= 30 kg/m2 or <= 16 kg/m2
* Previously known other malignancies
* Second primary cancer
* Previously received chemotherapy or radiotherapy
* Severe malnutrition with administration of TPN is indicated
* Pregnancy or lactation
* CKD stage 4-5

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Percent weight change | 12 weeks
  The change of body weight (%) before and after chemotherapy treatment

SECONDARY OUTCOMES:
EORTC QLQ-C30 | 12 weeks
  The change of Global Quality of life before and after chemotherapy treatment score
Patient interpretation of the Patient-Generated Subjective Global Assessment | 12 weeks
  PG-SGA
EORTC QLQ-BR23 | 12 weeks
  The change of Global Quality of life before and after chemotherapy treatment score

CONTACTS AND LOCATIONS:
Overall Officials: Piyawan Tienchaiananda, Study Director — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Due to this study is performed on single institution. The study protocol will be provided later on published article.

REFERENCES:
- [Background] Muscaritoli M, Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Oldervoll L, Ravasco P, Solheim TS, Strasser F, de van der Schueren M, Preiser JC, Bischoff SC. ESPEN practical guideline: Clinical Nutrition in cancer. Clin Nutr. 2021 May;40(5):2898-2913. doi: 10.1016/j.clnu.2021.02.005. Epub 2021 Mar 15. PMID 33946039
- [Background] Hebuterne X, Lemarie E, Michallet M, de Montreuil CB, Schneider SM, Goldwasser F. Prevalence of malnutrition and current use of nutrition support in patients with cancer. JPEN J Parenter Enteral Nutr. 2014 Feb;38(2):196-204. doi: 10.1177/0148607113502674. PMID 24748626
- [Background] Dewys WD, Begg C, Lavin PT, Band PR, Bennett JM, Bertino JR, Cohen MH, Douglass HO Jr, Engstrom PF, Ezdinli EZ, Horton J, Johnson GJ, Moertel CG, Oken MM, Perlia C, Rosenbaum C, Silverstein MN, Skeel RT, Sponzo RW, Tormey DC. Prognostic effect of weight loss prior to chemotherapy in cancer patients. Eastern Cooperative Oncology Group. Am J Med. 1980 Oct;69(4):491-7. doi: 10.1016/s0149-2918(05)80001-3. PMID 7424938
- [Background] Sukaraphat N, Chewaskulyong B, Buranapin S. Dietary Counseling Outcomes in Locally Advanced Unresectable or Metastatic Cancer Patients Undergoing Chemotherapy. J Med Assoc Thai. 2016 Dec;99(12):1283-90. PMID 29952503
- [Background] Ovesen L, Allingstrup L, Hannibal J, Mortensen EL, Hansen OP. Effect of dietary counseling on food intake, body weight, response rate, survival, and quality of life in cancer patients undergoing chemotherapy: a prospective, randomized study. J Clin Oncol. 1993 Oct;11(10):2043-9. doi: 10.1200/JCO.1993.11.10.2043. PMID 8410128
- [Derived] Tienchaiananda P, Juntong M, Pintasiri P, Sa-Nguansai S, Payapwattanawong S, Maneenil K. Body weight change in a medical supplement group in patients with early breast cancer during chemotherapy: a randomized, controlled trial. Support Care Cancer. 2025 Mar 19;33(4):299. doi: 10.1007/s00520-025-09359-z. PMID 40106001